CLINICAL TRIAL: NCT00176683
Title: Assessing the Use of Capnography as a Guide for Endotracheal Intubation
Brief Title: The Use of Capnography as a Guide for Oral Intubation
Status: Terminated | Type: Observational
Why Stopped: study was suspended because of difficluty maintaining equipment
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: 0120010351
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Measurement
Keywords: intubation; capnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All comers: capnography used for all consenting subjects
  Interventions: Procedure: Capnography

INTERVENTIONS:
Procedure: Capnography — device which measures carbon dioxide at intubation

SUMMARY:
The purpose of this study is to assess if capnography can be utilized to assist in the process of endotracheal intubation; specifically, in locating the glottic opening. Ultimately this would result in a new use of capnography to aid in securing normal and difficult airways. Currently capnography is only utilized for the confirmation of endotracheal tube placement.

If successful, this study will provide information, and allow for the development of instrumentation that will assist in difficult airway management; specifically, in locating the glottic opening when visualization may be impaired. Ultimately, this technique will be useful for routine and emergency airway management.

DETAILED DESCRIPTION:
The purpose of this study is to assess if capnography can be utilized in the process of endotracheal intubation; specifically, in locating the glottic opening. Ultimately this would result in a new use of capnography to aid in securing normal and difficult airways. Currently capnography is only utilized for the confirmation of endotracheal tube placement.

If successful, this study will provide information, and allow for the development of instrumentation that will assist in difficult airway management; specifically, in locating the glottic opening when visualization may be impaired. Ultimately this technique will be useful for routine and emergency airway management.

ELIGIBILITY:
Inclusion Criteria:

* Patients for elective surgery, requiring general endotracheal anesthesia

Exclusion Criteria:

* Patients with a known or suspected difficult intubation
* Patients requiring specialized endotracheal tubes
* Patients with a history of tracheostomy
* Airway tumor or airway pathology

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving general anesthesia and requiring endotracheal intubation.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2005-07; Primary Completion 2008-09 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
successful intubation | at intubation

CONTACTS AND LOCATIONS:
Overall Officials: Glen Atlas, MD, Msc, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- New Jersey Medical School, Newark, New Jersey, United States